CLINICAL TRIAL: NCT05245006
Title: A First-in-Human, Pilot PET Imaging Study of 89Zr-DFO-YS5, an immunoPET Agent for Detecting CD46 Positive Malignancy in Men With Prostate Cancer
Brief Title: PET Imaging Study of 89Zr-DFO-YS5 in Men With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Flavell, MD, PhD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Fortis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Robert Flavell, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 209210; NCI-2022-01310 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: First-in-Human; immunoPET agent; CD46 positive malignancy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: 89Zr-DFO-YS5 (Experimental): Participants receive one dose of 89Zr-DFO-YS5 up to 3 millicurie (mCi), and undergo a whole body PET performed at 1-4 hours, approximately 20-28 hours, 48-96 hours, and 120-168 hours post injection for up to 4 scans total. The optimized scan time will be used for imaging in cohorts B and C. Participants have the option to receive a repeat 89Zr-DFO-YS5 PET at the time of disease progression.
  Interventions: Drug: 89Zr-DFO-YS5; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI)
- Cohort B: 89Zr-DFO-YS5, YS5 antibody (Experimental): Participants receive either a 20mg or 50mg dose of YS5 prior to imaging and administration of one dose of up to 3 millicurie (mCi) 89Zr-DFO-YS5 and then complete a single whole body PET scan at the optimal time determined in Cohort A. The optimal dose of unmodified YS5 antibody will be used in the following cohorts C & D. Participants have the option to receive a repeat 89Zr-DFO-YS5 PET at the time of disease progression.
  Interventions: Drug: 89Zr-DFO-YS5; Biological: YS5 antibody; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI)
- Cohort C: 89Zr-DFO-YS5, Optimal dose YS5 antibody (Experimental): Participants receive optimal dose of YS5 antibody prior to imaging and administration of one dose of up to 3 millicurie (mCi) 89Zr-DFO-YS5 and then complete a single whole body PET scan at the optimal time determined in Cohort A. Participants have the option to receive a repeat 89Zr-DFO-YS5 PET at the time of disease progression.
  Interventions: Drug: 89Zr-DFO-YS5; Biological: YS5 antibody; Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT); Procedure: Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: 89Zr-DFO-YS5 — 3 mCi will be administered intravenously
  Other Names: immunoPET agent; Imaging Agent
Biological: YS5 antibody — 20 or 50 mg administered intravenously
  Other Names: YS5; Unmodified YS5 antibody
  Arms: Cohort B: 89Zr-DFO-YS5, YS5 antibody; Cohort C: 89Zr-DFO-YS5, Optimal dose YS5 antibody
Procedure: Positron Emission Tomography (PET)/Computerized tomography (CT) — Imaging which combines a CT scan and a PET scan
  Other Names: PET/CT; PET/CT Scan; Whole Body PET/CT
Procedure: Positron Emission Tomography (PET)/Magnetic Resonance Imaging (MRI) — Imaging which combines an MRI scan and a PET scan
  Other Names: PET/CT; PET/MRI Scan; Whole Body PET/MRI

SUMMARY:
CD46 is an exciting new therapeutic target in prostate cancer, with the antibody drug conjugate FOR46 under investigation in phase I clinical trials. The hypothesis of the study is that CD46 expression, measured via our novel imaging biomarker, is a characteristic feature of mCRPC, and particularly common in the most lethal forms of the disease including adenocarcinoma and Small-cell neuroendocrine carcinoma (SCNC). These data will provide crucial information about the feasibility of targeting cluster of differentiation 46 (CD46) in mCRPC, will be used guide the development of novel therapeutic and theranostic agents, to help develop treatments that improve outcomes for men with the most lethal forms of prostate cancer.

DETAILED DESCRIPTION:
This single center imaging study involves one microdose of the imaging agent, followed by whole body PET imaging. Imaging data will be acquired in up to four PET studies to determine tumor and normal tissue uptake and dosimetry.

PRIMARY OBJECTIVES:

1. To determine the optimal time point for imaging (based on analyzing the 4 scans of all participants using 89Zr-DFO-YS5 PET post-injection). (Cohort A)
2. To determine the optimal antibody dose for imaging using 89Zr-DFO-YS5 PET. (Cohort B).
3. To determine the sensitivity of metastatic lesion detection in mCRPC using 89Zr-DFO-YS5 PET as compared with conventional imaging (Cohorts C)

SECONDARY OBJECTIVES:

1. To determine the safety of 89Zr-DFO-YS5.
2. To determine average organ uptake of 89Zr-DFO-YS5 (Cohort C).
3. To descriptively report the patterns of intra-tumoral uptake of 89Zr-DFO-YS5 on whole body PET, including by site of disease, uptake by tumor type, inter-tumoral and inter-patient heterogeneity, and tumor-to-background signal (Cohorts C).

OUTLINE: Participants were originally assigned to 1 of 3 cohorts. Cohort B is closed to accrual. Enrollment into Cohort A and C are ongoing.

Cohort A: PET imaging data will be acquired up to four times to determine tumor and normal tissue uptake and dosimetry. The optimized scan time will be used for imaging in Cohorts B and C.

(CLOSED) Cohort B: A dose of cold, non-radiolabeled antibody administered will be varied to determine the optimal antibody dose for image quality. The optimized antibody dose will be used in Cohort C. Participants will be followed for an additional 4-5 weeks after dose administration to assess for adverse events.

Cohort C: PET imaging will be acquired at the optimal time point and optimal antibody dose determined in Cohorts A & B, and have the option to obtain an repeat scan at the time of disease progression.

All participants will be followed for up to 5 weeks after their first scan to assess for adverse events and will be followed-up until progression. At the time of progression, participants will have the option to receive a repeat scan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed metastatic, castration resistant prostate cancer (mCRPC).
2. Age >=18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky >60%).
4. Demonstrates adequate organ function as defined below:

   1. Total bilirubin <1.5 X upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase (SGOT)) <= 3 X institutional upper limit of normal (ULN).
   3. Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) <= 3 X institutional ULN.
   4. Serum creatinine <=1,5 X institutional ULN or calculated creatinine clearance (Glomerular filtration rate (GFR)) >= 60 mL/min, calculated using the Cockcroft-Gault equation.
5. Ability to understand a written informed consent document, and the willingness to sign it.
6. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Patients who because of age, general medical, or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal time point for imaging using 89Zr-DFO-YS5 PET post-injection (Cohort A) | Up to 7 days
  For Cohort A, the optimal time point will be selected based on optimal maximun Standardized uptake value (SUVmax) of metastatic lesions, and ratio of SUVmax to blood pool. Due to the limited samples, the investigator will use all available lesions without considering the location of the lesions or the possible intra-correlation of the lesions from the same participant.
Optimal antibody dose for imaging using 89Zr-DFO-YS5 PET (Cohort B) | Up to 7 days
  For Cohort B, the optimal dose of antibody will be selected based on the optimal SUVmax of metastatic lesions, and ratio of SUVmax to blood pool. Due to the limited samples, the investigator will use all available lesions without considering the location of the lesions or the possible intra-correlation of the lesions from the same participant.
Proportion of participants with metastatic lesions accurately detected in mCRPC using 89Zr-DFO-YS5 PET (sensitivity) (Cohort C) | Up to 24 months
  Sensitivity is the probability that a test will indicate disease among those with the actual disease: True Positive / (True Positive + False Negative). Lesions will be graded on a semi-quantitative scale ranging from 1-5 as is common for 89Zr-antibody human imaging studies (1 = no uptake, 2 = probably no uptake, 3 = equivocal, 4 = probably positive, 5 = definitely positive). Using as a cut-off to 4 or 5 on the semi-quantitative scale, the sensitivity of 89Zr-DFO-YS5 PET will be descriptively reported on a lesion-per-lesion basis, using as reference standard staging scans including CT or MRI of the chest/abdomen/pelvis and whole body bone scan. The sensitivity estimate will be based on lesion level without considering the location of the lesions or the possible intra-correlation of the lesions from the same patient.
Median SUVmax (Cohort C) | Up to 24 months
  The median and range of SUVmax across all metastatic lesions per participant will be descriptively reported using mediastinal blood pool and normal organ as background uptake values will be reported with range of SUVmax.
Average SUVmax (SUVmax-ave) (Cohort C) | Up to 24 months
  The average SUVmax-ave across all metastatic lesions per participant will be descriptively reported using mediastinal blood pool and normal organ as background uptake values for all cohorts will be reported with 95% confidence intervals

SECONDARY OUTCOMES:
Proportion of participants with treatment-related Adverse Events | Up to 3 weeks after last dose administration, approximately 35 days
  The frequency and severity of adverse events following Zr-DFO-YS5 injection will be descriptively reported, using CTCAE version 5.0
Average organ uptake of 89Zr-DFO-YS5 (Cohort C) | Up to 24 months
  Average organ uptake of 89Zr-DFO-YS5 on PET will be estimated.
Intra-tumoral uptake of 89Zr-DFO-YS5 by tumor type (Cohort C) | Up to 24 months
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported
Intra-tumoral uptake of 89Zr-DFO-YS5 by Site of Disease (Cohort C) | Up to 24 months
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported
Inter-tumoral heterogeneity (Cohort C) | Up to 24 months
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported to assess for Inter-tumoral heterogeneity.
Inter-participant heterogeneity (Cohort C) | Up to 24 months
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported to assess for Inter-participant heterogeneity
Tumor-to-background signal (Cohort C) | Up to 24 months
  The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No